CLINICAL TRIAL: NCT02714036
Title: A Multi-Center, Open-Label Biomarker Study to Evaluate MN-166 in Subjects With Amyotrophic Literal Sclerosis (ALS)
Brief Title: A Biomarker Study to Evaluate MN-166 in Subjects With Amyotrophic Literal Sclerosis (ALS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Collaborators: Massachusetts General Hospital (Other); South Shore Neurologic Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MN-166-ALS-1202
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ibudilast

STUDY DESIGN:
Masking Description: Participants were assigned to one of 2 groups at the discretion of the Principal Investigator.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular (Experimental): Participants will receive up to 100 mg /day MN-166 for 36 weeks. MN-166 dosing may vary based on individual tolerability.
  Interventions: Drug: ibudilast
- Flexible (Experimental): Participants will receive up to 100 mg /day MN-166 for 36 weeks. MN-166 dosing may vary based on individual tolerability. Participants will have all assessments except PET scans.
  Interventions: Drug: Ibudilast

INTERVENTIONS:
Drug: ibudilast — Ibudilast is a small molecule that crosses the blood-brain barrier after oral administration. Its potential as a neuroprotective agent is based on in vitro and in vivo evidence of its ability to reduce microglial activation, inhibit microglia-monocyte recruitment to the central nervous system (CNS), and trigger the release of neurotrophic factors.
  Other Names: MN-166
  Arms: Regular
Drug: Ibudilast — Ibudilast is a small molecule that crosses the blood-brain barrier after oral administration. Its potential as a neuroprotective agent is based on in vitro and in vivo evidence of its ability to reduce microglial activation, inhibit microglia-monocyte recruitment to the central nervous system (CNS), and trigger the release of neurotrophic factors.
  Other Names: MN-166
  Arms: Flexible

SUMMARY:
This is a multi-center, open-label study of MN-166 (ibudilast) in subjects with ALS. To be eligible subjects must meet the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS. Safety, tolerability, blood, neuro-imaging biomarkers, and clinical outcomes will be collected on all subjects. Subjects will receive study drug for 36 weeks.

The study will consist of a Screening Phase (up to 6 weeks), an Open-Label Treatment Phase (36 weeks) and an Off-Treatment Follow-up Phase (4 Weeks).

Number of Subjects (Planned):

Approximately 45 subjects are planned to be screened with the goal of enrolling 35 subjects.

DETAILED DESCRIPTION:
This is a multi-center, open-label study of MN-166 (ibudilast) in subjects with ALS. To be eligible subjects must meet the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS. Safety, tolerability, blood, neuro-imaging biomarkers, and clinical outcomes will be collected on all subjects. Subjects will receive study drug for 36 weeks.

The study will consist of a Screening Phase (up to 6 weeks), an Open-Label Treatment Phase (36 weeks) and a Off-Treatment Follow-up Phase (4 Weeks).

During the Screening Phase, eligible ALS subjects will sign an informed consent form and the following screening assessments will be performed: review of inclusion/exclusion criteria: El Escorial ALS Diagnostic criteria, medical history and demographics, ALS diagnosis history, physical and neurological examination, U. Penn upper motor Neuron Burden (UMNB), pulmonary function tests, vital signs including height and weight, blood for safety labs including TSPO affinity test, ECG and review and documentation of concomitant medications and therapies.

Screening Phase (up to 6 weeks) The Treatment Phase will consist of a Baseline visit and 3 subsequent clinic visits at Weeks 4, 12, 24, and 36. Telephone follow-ups will occur at Weeks 1, 2, 8, 16, 20, 28, and 32.

Open-Label Treatment Phase (36 weeks) At the Baseline visit, subjects will return to the clinic and the following assessments will be performed/administered: review of inclusion and exclusion criteria for continued eligibility, vital signs, blood for safety labs and biomarkers, ECG, ALSFRS-R questionnaire, slow vital capacity (SVC), baseline strength as measured by hand held dynamometry (HHD), and Columbia Suicide Severity Rating Scale (C-SSRS). At this visit, study drug will be dispensed, and adverse events, concomitant medications and therapies will be assessed and documented. At subsequent visits during the Treatment Phase, similar assessments will be performed.

In addition, a [11C]PBR28-PET scan will be performed once between the Screening and Baseline visit, and once between the Week 12 and Week 28 phone calls. The ALSFRS-R, SVC and U Penn Upper Motor Neuron Burden will be repeated on the same day as the PET scans.

The follow-up visit will consist of a telephone call to document adverse events and concomitant therapies

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed as having possible, probable, probable-laboratory supported, or definite ALS, either sporadic or familial according to modified El Escorial criteria.
2. Age 18 or above, able to provide informed consent, and safely comply with study procedures.
3. Vital capacity (VC) of at least 50% predicted value for gender, height and age at screening visit, or in the opinion of the study physician, able to safely tolerate study procedures. (Not applicable to flexible arm)
4. Subject must be able to swallow oral medication at the Baseline Visit and expected to be able to swallow the capsules throughout the course of the study.
5. Subject must not have taken riluzole for at least 30 days or be on a stable dose of riluzole for at least 30 days, prior to screening (riluzole-naïve participants are permitted in the study). (Not applicable to flexible arm)
6. Women must not be able to become pregnant (e.g. post-menopausal, surgically sterile, or using adequate birth control) for the duration of the study and 3 months after study completion.
7. Males should practice contraception for the duration of the study and 3 months after completion.
8. Ability to safely lie flat for 90 min for PET procedures in the opinion of the study physician. (Not applicable to flexible arm)
9. High or mixed affinity to bind TSPO protein (Ala/Ala or Ala/Thr) (not applicable to flexible arm).
10. Upper motor Neuron Burden (UMNB) Score ≥25 (out of 45) at screening visit. (Not applicable to flexible arm)

Exclusion Criteria:

1. Abnormal liver function defined as AST and/or ALT > 3 times the upper limit of the normal.
2. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal.
3. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the participant to provide informed consent, according to PI judgment.
4. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant if they were to participate in the study.
5. History of HIV, clinically significant chronic hepatitis, or other active infection.
6. Active inflammatory condition of autoimmune disorder (Not applicable to flexible arm)
7. Females must not be lactating or pregnant.
8. Active participation in another ALS clinical trial or exposure to an off-label ALS experimental treatment within 30 days of the Baseline Visit (Not applicable to flexible arm)
9. Exposure to immunomodulatory medications within 30 days of the Baseline Visit. (Not applicable to flexible arm)
10. Any contraindication to undergo MRI studies such as

    * History of a cardiac pacemaker or pacemaker wires
    * Metallic particles in the body
    * Vascular clips in the head
    * Prosthetic heart valves
    * Claustrophobia (Not applicable to flexible arm)
11. Radiation exposure that exceeds the site's current guidelines (Not applicable to flexible arm)
12. EKG finding of QTc prolongation > 450 msec for males and > 470 msec for females at screening or baseline.
13. Not on any prohibitive medication or known QT prolonging medication:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suma Babu, MBBS, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - South Shore Neurologic Associates, P.C., Patchogue, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Chalabi A, Hardiman O. The epidemiology of ALS: a conspiracy of genes, environment and time. Nat Rev Neurol. 2013 Nov;9(11):617-28. doi: 10.1038/nrneurol.2013.203. Epub 2013 Oct 15. PMID 24126629
- [Background] Chio A, Logroscino G, Hardiman O, Swingler R, Mitchell D, Beghi E, Traynor BG; Eurals Consortium. Prognostic factors in ALS: A critical review. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):310-23. doi: 10.3109/17482960802566824. PMID 19922118
- [Background] Chio A, Logroscino G, Traynor BJ, Collins J, Simeone JC, Goldstein LA, White LA. Global epidemiology of amyotrophic lateral sclerosis: a systematic review of the published literature. Neuroepidemiology. 2013;41(2):118-30. doi: 10.1159/000351153. Epub 2013 Jul 11. PMID 23860588
- [Background] Turner MR, Hardiman O, Benatar M, Brooks BR, Chio A, de Carvalho M, Ince PG, Lin C, Miller RG, Mitsumoto H, Nicholson G, Ravits J, Shaw PJ, Swash M, Talbot K, Traynor BJ, Van den Berg LH, Veldink JH, Vucic S, Kiernan MC. Controversies and priorities in amyotrophic lateral sclerosis. Lancet Neurol. 2013 Mar;12(3):310-22. doi: 10.1016/S1474-4422(13)70036-X. PMID 23415570
- [Background] Miller RG, Mitchell JD, Moore DH. Riluzole for amyotrophic lateral sclerosis (ALS)/motor neuron disease (MND). Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD001447. doi: 10.1002/14651858.CD001447.pub3. PMID 22419278
- [Background] Henkel JS, Beers DR, Siklos L, Appel SH. The chemokine MCP-1 and the dendritic and myeloid cells it attracts are increased in the mSOD1 mouse model of ALS. Mol Cell Neurosci. 2006 Mar;31(3):427-37. doi: 10.1016/j.mcn.2005.10.016. Epub 2005 Dec 5. PMID 16337133
- [Background] Boillee S, Yamanaka K, Lobsiger CS, Copeland NG, Jenkins NA, Kassiotis G, Kollias G, Cleveland DW. Onset and progression in inherited ALS determined by motor neurons and microglia. Science. 2006 Jun 2;312(5778):1389-92. doi: 10.1126/science.1123511. PMID 16741123
- [Background] Butovsky O, Siddiqui S, Gabriely G, Lanser AJ, Dake B, Murugaiyan G, Doykan CE, Wu PM, Gali RR, Iyer LK, Lawson R, Berry J, Krichevsky AM, Cudkowicz ME, Weiner HL. Modulating inflammatory monocytes with a unique microRNA gene signature ameliorates murine ALS. J Clin Invest. 2012 Sep;122(9):3063-87. doi: 10.1172/JCI62636. Epub 2012 Aug 6. PMID 22863620
- [Background] Koval ED, Shaner C, Zhang P, du Maine X, Fischer K, Tay J, Chau BN, Wu GF, Miller TM. Method for widespread microRNA-155 inhibition prolongs survival in ALS-model mice. Hum Mol Genet. 2013 Oct 15;22(20):4127-35. doi: 10.1093/hmg/ddt261. Epub 2013 Jun 4. PMID 23740943
- [Background] Brettschneider J, Del Tredici K, Toledo JB, Robinson JL, Irwin DJ, Grossman M, Suh E, Van Deerlin VM, Wood EM, Baek Y, Kwong L, Lee EB, Elman L, McCluskey L, Fang L, Feldengut S, Ludolph AC, Lee VM, Braak H, Trojanowski JQ. Stages of pTDP-43 pathology in amyotrophic lateral sclerosis. Ann Neurol. 2013 Jul;74(1):20-38. doi: 10.1002/ana.23937. Epub 2013 Jun 19. PMID 23686809
- [Background] Henkel JS, Engelhardt JI, Siklos L, Simpson EP, Kim SH, Pan T, Goodman JC, Siddique T, Beers DR, Appel SH. Presence of dendritic cells, MCP-1, and activated microglia/macrophages in amyotrophic lateral sclerosis spinal cord tissue. Ann Neurol. 2004 Feb;55(2):221-35. doi: 10.1002/ana.10805. PMID 14755726
- [Background] Kuhle J, Lindberg RL, Regeniter A, Mehling M, Steck AJ, Kappos L, Czaplinski A. Increased levels of inflammatory chemokines in amyotrophic lateral sclerosis. Eur J Neurol. 2009 Jun;16(6):771-4. doi: 10.1111/j.1468-1331.2009.02560.x. Epub 2009 Feb 19. PMID 19236470
- [Background] Moreau C, Devos D, Brunaud-Danel V, Defebvre L, Perez T, Destee A, Tonnel AB, Lassalle P, Just N. Elevated IL-6 and TNF-alpha levels in patients with ALS: inflammation or hypoxia? Neurology. 2005 Dec 27;65(12):1958-60. doi: 10.1212/01.wnl.0000188907.97339.76. PMID 16380619
- [Background] Zurcher NR, Loggia ML, Lawson R, Chonde DB, Izquierdo-Garcia D, Yasek JE, Akeju O, Catana C, Rosen BR, Cudkowicz ME, Hooker JM, Atassi N. Increased in vivo glial activation in patients with amyotrophic lateral sclerosis: assessed with [(11)C]-PBR28. Neuroimage Clin. 2015 Jan 19;7:409-14. doi: 10.1016/j.nicl.2015.01.009. eCollection 2015. PMID 25685708
- [Background] Sanftner LM, Gibbons JA, Gross MI, Suzuki BM, Gaeta FC, Johnson KW. Cross-species comparisons of the pharmacokinetics of ibudilast. Xenobiotica. 2009 Dec;39(12):964-77. doi: 10.3109/00498250903254340. PMID 19925385
- [Background] Cho Y, Crichlow GV, Vermeire JJ, Leng L, Du X, Hodsdon ME, Bucala R, Cappello M, Gross M, Gaeta F, Johnson K, Lolis EJ. Allosteric inhibition of macrophage migration inhibitory factor revealed by ibudilast. Proc Natl Acad Sci U S A. 2010 Jun 22;107(25):11313-8. doi: 10.1073/pnas.1002716107. Epub 2010 Jun 8. PMID 20534506
- [Background] Cox GM, Kithcart AP, Pitt D, Guan Z, Alexander J, Williams JL, Shawler T, Dagia NM, Popovich PG, Satoskar AR, Whitacre CC. Macrophage migration inhibitory factor potentiates autoimmune-mediated neuroinflammation. J Immunol. 2013 Aug 1;191(3):1043-54. doi: 10.4049/jimmunol.1200485. Epub 2013 Jun 24. PMID 23797673
- [Background] Wakita H, Tomimoto H, Akiguchi I, Lin JX, Ihara M, Ohtani R, Shibata M. Ibudilast, a phosphodiesterase inhibitor, protects against white matter damage under chronic cerebral hypoperfusion in the rat. Brain Res. 2003 Nov 28;992(1):53-9. doi: 10.1016/j.brainres.2003.08.028. PMID 14604772
- [Background] Suzumura A, Ito A, Yoshikawa M, Sawada M. Ibudilast suppresses TNFalpha production by glial cells functioning mainly as type III phosphodiesterase inhibitor in the CNS. Brain Res. 1999 Aug 7;837(1-2):203-12. doi: 10.1016/s0006-8993(99)01666-2. PMID 10434004
- [Background] Mizuno T, Kurotani T, Komatsu Y, Kawanokuchi J, Kato H, Mitsuma N, Suzumura A. Neuroprotective role of phosphodiesterase inhibitor ibudilast on neuronal cell death induced by activated microglia. Neuropharmacology. 2004 Mar;46(3):404-11. doi: 10.1016/j.neuropharm.2003.09.009. PMID 14975696
- [Background] Kiebala M, Maggirwar SB. Ibudilast, a pharmacologic phosphodiesterase inhibitor, prevents human immunodeficiency virus-1 Tat-mediated activation of microglial cells. PLoS One. 2011 Apr 8;6(4):e18633. doi: 10.1371/journal.pone.0018633. PMID 21494611
- [Background] Kagitani-Shimono K, Mohri I, Fujitani Y, Suzuki K, Ozono K, Urade Y, Taniike M. Anti-inflammatory therapy by ibudilast, a phosphodiesterase inhibitor, in demyelination of twitcher, a genetic demyelination model. J Neuroinflammation. 2005 Apr 6;2(1):10. doi: 10.1186/1742-2094-2-10. PMID 15813970
- [Background] Fujimoto T, Sakoda S, Fujimura H, Yanagihara T. Ibudilast, a phosphodiesterase inhibitor, ameliorates experimental autoimmune encephalomyelitis in Dark August rats. J Neuroimmunol. 1999 Mar 1;95(1-2):35-42. doi: 10.1016/s0165-5728(98)00251-3. PMID 10229113
- [Background] Barkhof F, Hulst HE, Drulovic J, Uitdehaag BM, Matsuda K, Landin R; MN166-001 Investigators. Ibudilast in relapsing-remitting multiple sclerosis: a neuroprotectant? Neurology. 2010 Mar 30;74(13):1033-40. doi: 10.1212/WNL.0b013e3181d7d651. Epub 2010 Mar 3. PMID 20200338
- [Background] Gibson LC, Hastings SF, McPhee I, Clayton RA, Darroch CE, Mackenzie A, Mackenzie FL, Nagasawa M, Stevens PA, Mackenzie SJ. The inhibitory profile of Ibudilast against the human phosphodiesterase enzyme family. Eur J Pharmacol. 2006 May 24;538(1-3):39-42. doi: 10.1016/j.ejphar.2006.02.053. Epub 2006 Mar 13. PMID 16674936
- [Background] Tominaga Y, Nakamura Y, Tsuji K, Shibata T, Kataoka K. Ibudilast protects against neuronal damage induced by glutamate in cultured hippocampal neurons. Clin Exp Pharmacol Physiol. 1996 Jun-Jul;23(6-7):519-23. doi: 10.1111/j.1440-1681.1996.tb02772.x. PMID 8800577
- [Background] Takuma K, Lee E, Enomoto R, Mori K, Baba A, Matsuda T. Ibudilast attenuates astrocyte apoptosis via cyclic GMP signalling pathway in an in vitro reperfusion model. Br J Pharmacol. 2001 Jul;133(6):841-8. doi: 10.1038/sj.bjp.0704146. PMID 11454657
- [Background] Yoshioka A, Shimizu Y, Hirose G, Kitasato H, Pleasure D. Cyclic AMP-elevating agents prevent oligodendroglial excitotoxicity. J Neurochem. 1998 Jun;70(6):2416-23. doi: 10.1046/j.1471-4159.1998.70062416.x. PMID 9603206
- [Background] Fox RJ. Primary neuroprotection: the Holy Grail of multiple sclerosis therapy. Neurology. 2010 Mar 30;74(13):1018-9. doi: 10.1212/WNL.0b013e3181d6b165. Epub 2010 Mar 3. No abstract available. PMID 20200341
- [Background] Owen DR, Yeo AJ, Gunn RN, Song K, Wadsworth G, Lewis A, Rhodes C, Pulford DJ, Bennacef I, Parker CA, StJean PL, Cardon LR, Mooser VE, Matthews PM, Rabiner EA, Rubio JP. An 18-kDa translocator protein (TSPO) polymorphism explains differences in binding affinity of the PET radioligand PBR28. J Cereb Blood Flow Metab. 2012 Jan;32(1):1-5. doi: 10.1038/jcbfm.2011.147. Epub 2011 Oct 19. PMID 22008728
- [Background] Kreisl WC, Jenko KJ, Hines CS, Lyoo CH, Corona W, Morse CL, Zoghbi SS, Hyde T, Kleinman JE, Pike VW, McMahon FJ, Innis RB; Biomarkers Consortium PET Radioligand Project Team. A genetic polymorphism for translocator protein 18 kDa affects both in vitro and in vivo radioligand binding in human brain to this putative biomarker of neuroinflammation. J Cereb Blood Flow Metab. 2013 Jan;33(1):53-8. doi: 10.1038/jcbfm.2012.131. Epub 2012 Sep 12. PMID 22968319
- [Background] Butovsky O, Jedrychowski MP, Cialic R, Krasemann S, Murugaiyan G, Fanek Z, Greco DJ, Wu PM, Doykan CE, Kiner O, Lawson RJ, Frosch MP, Pochet N, Fatimy RE, Krichevsky AM, Gygi SP, Lassmann H, Berry J, Cudkowicz ME, Weiner HL. Targeting miR-155 restores abnormal microglia and attenuates disease in SOD1 mice. Ann Neurol. 2015 Jan;77(1):75-99. doi: 10.1002/ana.24304. Epub 2014 Nov 27. PMID 25381879
- [Derived] Babu S, Hightower BG, Chan J, Zurcher NR, Kivisakk P, Tseng CJ, Sanders DL, Robichaud A, Banno H, Evora A, Ashokkumar A, Pothier L, Paganoni S, Chew S, Dojillo J, Matsuda K, Gudesblatt M, Berry JD, Cudkowicz ME, Hooker JM, Atassi N. Ibudilast (MN-166) in amyotrophic lateral sclerosis- an open label, safety and pharmacodynamic trial. Neuroimage Clin. 2021;30:102672. doi: 10.1016/j.nicl.2021.102672. Epub 2021 Apr 15. PMID 34016561

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analysis Sets:
  Safety (n=35, n=30 Regular arm, n=5 Flexible arm) = All participants initiated at least the first MN-166 dose.
  Intent-to-Treat (ITT) (n=30) = All participants initiated at least the first MN-166 dose, excluding Flexible arm.
  Modified ITT (n=22) = Subset of ITT who completed pre- and post-treatment PET scans.
  Per Protocol (PP) (n=16) Subset of ITT who successfully titrated up to and maintained the full dose of 50 mg bid.
Period: Overall Study
Arm/Group | Regular | Flexible
Started | 30 (Completed 36-week treatment and End of Study visit.) | 5
Completed | 18 | 1
Not Completed | 12 | 4
Not completed — Adverse Event | 9 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular | Flexible | Total
Number analyzed (Participants) | 30 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.3) | 54.0 (14.3) | 56.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 15
  Male | 16 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 5 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 5 | 35
Mean years since ALS onset [Mean (Full Range); unit: mean years since ALS onset] | 2.06 [0.4 to 5.9] | 1.93 [0.9 to 2.7] | 2.04 [0.4 to 5.9]
Mean delay between symptom onset and ALS diagnosis [Mean (Full Range); unit: Mean years] | 1.12 [0.0 to 4.6] | 0.74 [0.0 to 1.4] | 1.06 [0.0 to 4.6]
Site of ALS onset [Count of Participants; unit: Participants]
  Bulbar onset | 10 | 2 | 12
  Lower Limb | 9 | 2 | 11
  Upper Limb | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Impact of MN-166 on [11C]-PBR28 Uptake in the Motor Cortices and Brain Stem Measured by Positron Emission Tomography (PET) Imaging at 12 - 24 Weeks
Description: Glial activation will be estimated in eligible participants in the Regular arm by combined magnetic resonance positron emission tomography (MR-PET) using the [11C]-PBR28 radioligand. [11C]-PBR28 uptake is quantified as the ratio of the standardized uptake value (SUVR). An independent neuroimaging rater blinded to the clinical data will assess for quality control of the PBR28-PET images and SUVR. The primary analysis will be performed on the modified Intent-to-Treat (mITT) population. The median (90% confidence interval [CI]) changes from baseline in SUVR from pre- to post-treatment visit will be presented.
Time Frame: 12- 24 weeks (post treatment [11C]-PBR28-PET scan will be performed between the Week 12 and Week 24 visits.
Population: modified Intent-to-Treat population
Measure: Median (90% Confidence Interval); unit: SUV ratio
Arm/Group | Regular
Number analyzed (Participants) | 22
SUV ratio | 0.0015 [-0.0082 to 0.0205]

2. Primary Outcome: Impact of MN-166 on Several Markers of Neuro-inflammation Measured by Blood Biomarkers at Week 36
Description: Mean change from baseline (pre-dose) to Week 36 in blood biomarkers for neuroinflammation, including macrophage migration inhibitory factor (MIF), tumor necrosis factor (TNF)-alpha, and neurofilament light (NfL). All blood biomarkers are measured in picograms/milliliter (pg/mL).
Time Frame: 36 weeks
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: picograms/milliliters
Arm/Group | Regular
Number analyzed (Participants) | 30
picograms/milliliters
  macrophage migration inhibitory factor | -673387.22 (943313.53)
  tumor necrosis factor-alpha | -0.31 (0.57)
  neurofilament light | 21.43 (47.71)

3. Secondary Outcome: Safety and Tolerability of MN-166 Over 36 Weeks
Description: Clinical and laboratory treatment-emergent adverse events (TEAEs) will be collected and stratified by severity, persistence over time, and relationship to study drug.
Time Frame: 36 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Flexible: Participants will receive MN-166 up to 100 mg/day for 36 weeks. MN-166 dosing may vary based on individual tolerability. Participants will have all assessments except PET scans.
Arm/Group | Regular | Flexible
Number analyzed (Participants) | 30 | 5
Participants | 30 | 5

4. Secondary Outcome: Evaluate the Effect of MN-166 on ALS Clinical Outcomes (ALS Functional Rating Scale-revised [ALSFRS-R]) Over 36 Weeks.
Description: Mean change from baseline to Week 36 on ALSFRS-R score. ALSFRS-R rating scale is a tool to assess patient's capability and independence in 12 functional activities. The ALSFRS-R total score is a composite of sub-scores measuring speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing and hygiene, turning in bed and adjusting bed clothes, walking, climbing stairs, dyspnea, orthopnea, and respiratory insufficiency. Each subscale ranges from 0 (no ability) to 4 (normal ability). The ALSFRS-R score is the sum total ranging from 0 (zero) to 48, with higher scores meaning better outcome.
Time Frame: 36 weeks
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: Total ALSFRS-R score
Arm/Group | Regular
Number analyzed (Participants) | 30
Total ALSFRS-R score | -4.5 (4.5)

5. Secondary Outcome: Mean Change From Baseline in Slow Vital Capacity (Percent Predicted) Normal Volume at Week 36
Description: Slow vital capacity (SVC) is the maximum volume of air that can be slowly exhaled after slow, maximal inhalation, measured in liters. The maximum volume expired is converted to percent of predicted (% pred.) normal volume. Higher SVC (% pred.) normal volume indicates better pulmonary function. The results below reflect the mean change in SVC (% pred.) from baseline to week 36.
Time Frame: 36 weeks
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: percent predicted normal volume
Arm/Group | Regular
Number analyzed (Participants) | 30
percent predicted normal volume | -9.27 (11.23)

6. Secondary Outcome: Mean Change From Baseline in Isometric Strength as Measured by Hand-held Dynamometry (HHD) at Week 36.
Description: HHD assesses isometric strength using a MicroFET2 hand-held dynamometer in kilograms (kg). To calculate megascores, the mean and standard deviation of each muscle group, without regard to laterality, is calculated from the baseline assessment. Nine upper and lower extremity muscles or muscle groups were examined: shoulder flexion, elbow flexion, wrist extension, first dorsal interosseous contraction, hip flexion, knee extension, and ankle dorsiflexion. Each group was measured at least twice bilaterally and the average of the 2 highest measurements were analyzed. To calculate megascores, the mean and standard deviation of each group were calculated from baseline.
Time Frame: 36 weeks
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Regular
Number analyzed (Participants) | 30
kilograms
  upper limbs, proximal | -0.5803 (0.8108)
  upper limbs, distal | -0.5004 (0.4823)
  upper limbs, cumulated | -0.5324 (0.5738)
  lower limbs, proximal | -0.2778 (0.7749)
  lower limbs, distal | -0.3525 (0.6492)
  lower limbs, cumulated | -0.3151 (0.6824)
  cumulated | -0.4358 (0.5863)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Regular | Flexible
All-Cause Mortality (participants affected / at risk) | 2/30 | 0/5
Serious Adverse Events (participants affected / at risk) | 6/30 | 0/5
Other Adverse Events (participants affected / at risk) | 30/30 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regular (N=30) | Flexible (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe, not related to Ibudilast, not related to ALS. There was no action taken with the IP. The SAE resolved. Subject died.
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient no longer able to swallow food.
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Pulmonary embolism was assessed as life-threatening by intensity, not related to Ibudilast, not related to ALS. There was no action taken with the IP. Subject died.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Respiratory failure not related to Ibudilast, related to ALS. Treatment with Ibudilast was interrupted.
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regular (N=30) | Flexible (N=5)
nausea (Gastrointestinal disorders) | 13 (13) | 3 (3)
dysphagia (Gastrointestinal disorders) | 8 (8) | 0 (0)
diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
salivary hypersecretion (Gastrointestinal disorders) | 4 (4) | 2 (2)
abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1)
defecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 6 (6) | 1 (1)
dizziness (Nervous system disorders) | 6 (6) | 0 (0)
dysarthria (Nervous system disorders) | 3 (3) | 0 (0)
restless leg syndrome (Nervous system disorders) | 1 (1) | 1 (1)
slow speech (Nervous system disorders) | 2 (2) | 0 (0)
dysgeugia (Nervous system disorders) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 15 (15) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
stoma site erythema (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
fatigue (General disorders) | 11 (11) | 2 (2)
chest discomfort (General disorders) | 2 (2) | 0 (0)
edema peripheral (General disorders) | 2 (2) | 0 (0)
pain (General disorders) | 2 (2) | 0 (0)
disease progression (General disorders) | 0 (0) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
insomnia (Psychiatric disorders) | 5 (5) | 2 (2)
depressed mood (Psychiatric disorders) | 2 (2) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0)
oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hot flush (Vascular disorders) | 6 (6) | 0 (0)
deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 1 (1)
weight decreased (Investigations) | 4 (4) | 1 (1)
chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
urine odor abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT02714036/Prot_SAP_000.pdf